CLINICAL TRIAL: NCT06192147
Title: The Phenotype and Clinical Intervention of High Branched Chain Amino Acid Type of Polycystic Ovary Syndrome
Brief Title: The Phenotype and Clinical Intervention of High BCAA Type of PCOS
Acronym: BCAAPCOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Xiaoyu, Dr, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCAAPCOS20231219
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Accurate classification; High branched chain amino acids
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): On the basis of conventional treatment, a protein restricted diet combined with vitamin D intervention plan is given
  Interventions: Dietary Supplement: protein restricted diet combined with vitamin D intervention
- control group (No Intervention): basic conventional treatment

INTERVENTIONS:
Dietary Supplement: protein restricted diet combined with vitamin D intervention — On the basis of conventional treatment, a protein restricted diet combined with vitamin D intervention plan is given
  Arms: intervention group

SUMMARY:
Polycystic ovary syndrome is one of the main diseases leading to infertility in women of childbearing age. In addition to endocrine and reproductive dysfunction, it is often accompanied by significant metabolic abnormalities, which seriously affect long-term health and quality of life. Our preliminary research found that 68% of PCOS patients have significantly increased branched chain amino acid content, accompanied by a decrease in clinical pregnancy rate and an increase in miscarriage rate, which poses challenges to the diagnosis and treatment of PCOS. Based on this, we propose a new PCOS typing strategy that uses the concentration of branched chain amino acids as an evaluation indicator to diagnose high branched chain amino acid PCOS, where the serum BCAA concentration is higher than 405 μ Mol/L is diagnosed as high branched chain amino acid PCOS. According to the different degrees of elevation of branched chain amino acids, they are further divided into common type and ultra-high type, and the impact of different concentrations of branched chain amino acids on pregnancy outcomes, pregnancy complications, and newborns after assisted reproductive technology is analyzed; Based on the typical clinical and metabolic phenotypes of high branched chain amino acid type PCOS patients, corresponding intervention strategies are formulated. By analyzing the clinical pregnancy outcomes, pregnancy complications, and neonatal conditions of patients in the combination intervention group (protein restricted diet combined with vitamin D supplementation) and the conventional treatment group, safe and effective intervention methods are determined.

DETAILED DESCRIPTION:
Based on this, we propose a new PCOS typing strategy that uses the concentration of branched chain amino acids as an evaluation indicator to diagnose high branched chain amino acid PCOS, where the serum BCAA concentration is higher than 405 μ Mol/L is diagnosed as high branched chain amino acid PCOS. According to the different degrees of elevation of branched chain amino acids, they are further divided into common type and ultra-high type, and the impact of different concentrations of branched chain amino acids on pregnancy outcomes, pregnancy complications, and newborns after assisted reproductive technology is analyzed; Based on the typical clinical and metabolic phenotypes of high branched chain amino acid type PCOS patients, corresponding intervention strategies are formulated. By analyzing the clinical pregnancy outcomes, pregnancy complications, and neonatal conditions of patients in the combination intervention group (protein restricted diet combined with vitamin D supplementation) and the conventional treatment group, safe and effective intervention methods are determined.

ELIGIBILITY:
Inclusion Criteria:

The included population is PCOS patients who are seeking their first IVF treatment at the Reproductive Medicine Center of Peking University Third Hospital, aged 20-40 years old. PCOS diagnosis meets two of the following three criteria based on the 2003 Rotterdam criteria: clinical manifestations of oligomenorrhea and/or amenorrhea, hyperandrogenism or hyperandrogenism (hirsutism, acne, etc.), PCO like changes in the ovaries under ultrasound, while excluding diseases such as hyperprolactinemia, congenital adrenal hyperplasia, Cushing syndrome, and androgen secreting tumors. All selected subjects have no medical history of taking steroid drugs within 3 months.

Exclusion Criteria:

1) Refusing to sign informed consent or unable to follow up on time; 2) Severe complications requiring cessation of treatment (>2 weeks) or termination of treatment; 3) Patients should take vitamin D orally before enrollment (baseline data still needs to be recorded for later statistical analysis); 4) Any unstable or medical condition that affects patient safety and research compliance. 5) Male partners have severe male infertility factors; 6) Patients undergoing embryo analysis using pre implantation genetic testing techniques (PGT-A/SR/M).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | one year
  Clinical pregnancy patients/(transplant cycle) patients × 100%

SECONDARY OUTCOMES:
Excellent embryo rate | one year
  number of high-quality embryos/number of normal fertilized cleavage embryos × 100%
Fertilization rate | one year
  number of fertilized eggs/number of retrieved eggs × 100%
  Implantation rate=number of gestational sacs/total number of transplanted embryos × 100% (the number of gestational sacs in a single embryo transfer is only counted as 1)
Early miscarriage rate | one year
  number of natural abortion cycles within 12 weeks of pregnancy/number of clinical pregnancy cycles × 100%
Live birth rate (transplant cycle) | one year
  number of live births/number of transplant cycles × 100%
The incidence of pregnancy complications | one year
  number of pregnancy complications/number of clinical pregnancy cycles × 100%